CLINICAL TRIAL: NCT00065962
Title: Multisite Controlled Secretin Trial in Autism
Brief Title: Secretin for the Treatment of Autism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 5P01HD035465 (NIH); NICHD-23; 57-937; 5P01HD035465 (NIH); Supplement CRC99-3; 3P01HD035468 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Autism
Keywords: Pervasive Developmental Disorders; Secretin, synthetic porcine; Secretin, biological porcine; Autism Diagnostic Observation Schedule - Generic (ADOS-G); Rimland Questionnaire; Expressive Vocabulary Test; MacArthur Communication Inventory; Aberrant Behavior Checklist
MeSH Terms: conditions — Autistic Disorder; Child Development Disorders, Pervasive | interventions — Secretin

INTERVENTIONS:
Drug: secretin, synthetic porcine
Drug: secretin, biologically derived porcine

SUMMARY:
Many drugs used to treat autism target specific symptoms, such as hyperactivity and aggressiveness. Few drugs target the core autistic symptoms of impaired social interaction and communication. This study will evaluate two forms of the drug secretin for the treatment of core autistic symptoms.

DETAILED DESCRIPTION:
Autism is a disorder characterized by impairments of social interactions, verbal and nonverbal communication, and preoccupation with unusual activities or interests, particularly stereotyped or repetitive movements. This debilitating disorder is estimated to occur in 2 to 10 of every 10,000 births. A primary focus in pyschopharmacological intervention has been to treat specific associated symptoms, such as hyperactivity, aggressiveness, and temper tantrums; there are few pharmacologic treatments directed toward core autistic symptoms.

Secretin is a gut hormone with binding sites in the brain. Previous research has described three patients with autism who underwent diagnostic endoscopy for gastrointestinal complaints and experienced dramatic improvement in autistic symptoms following the administration of intravenous secretin given as part of endoscopy. Though the results of this single, uncontrolled study have limited interpretive value, many autistic children have been exposed and continue to be exposed to this potential treatment in an uncontrolled manner. This double blind, placebo-controlled trial will evaluate the safety and efficacy of secretin for the treatment of autism.

Participants will be randomly assigned to one of three treatment groups: synthetic porcine secretin (sPS), biologically derived porcine secretin (bPS), or placebo. Each participant will be given an initial intravenous dose of 0.1 ml of their assigned treatment at the appropriate dose (0.2 ug for sPS and 1 CU for bPS). If no allergic reaction occurs within one minute, the participants will continue in the study and receive the full remaining dose over one minute. Participants will be evaluated one week before and four weeks after infusion for social, communication, and behavioral functioning as measured by Autistic Diagnostic Observation Schedule Generic (by blinded raters); Rimland Questionnaires (by parents and teachers); Expressive Vocabulary Test; MacArthur Communication Inventory (by parents and teachers); and Aberrant Behavior Checklist (by parents and teachers). Participants will also have a physical exam and blood and urine tests. After completion of preliminary data analysis, placebo patients will be offered open label therapy if appropriate.

ELIGIBILITY:
Inclusion Criteria

* Autism based on DSM-IV criteria
* IQ > 35
* Medically fit for the study in the judgment of the study officials

Exclusion Criteria

* Prior administration of secretin
* Acute or chronic pancreatitis
* Use of anticholinergics within 72 hours of study entry or anticipated need for anticholinergics during study
* Allergies to pork products
* Use of investigational drug within 1 month of study entry
* Change in any medication or other therapeutic modality being used to treat any neurodevelopmental or gastrointestinal symptoms of the underlying autism disorder within 1 month of study entry
* Any medical condition which, in the judgment of the investigator, would make the patient unable to safely participate in the study or comply with all study procedures
* Any medical diagnosis which could account for autistic spectrum disorder (i.e., Rett syndrome, Fragile X, tuberous sclerosis, disintegrative disorder, epilepsy, Landau Kleffner, other mental retardation syndromes, or history of severe motor delays or current sensory or motor impairment such as cerebral palsy)
* Hearing or visual impairments
* Use of psychotropic medications (except for occasional symptomatic use for sleep, etc.) within 6 months of study entry

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 85
Dates: Start 1999-06; Study Completion 2000-05

CONTACTS AND LOCATIONS:
Overall Officials: Alan Unis, MD, Study Director — University of Washington; Geraldine Dawson, PhD, Principal Investigator — University of Washington; Edward Goldson, MD, Study Director — University of Colorado, Denver; Sally Rogers, PhD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Children's Hospital, Denver, Colorado
  - Center on Human Development and Disability, Seattle, Washington

REFERENCES:
- [Background] Unis AS, Munson JA, Rogers SJ, Goldson E, Osterling J, Gabriels R, Abbott RD, Dawson G. A randomized, double-blind, placebo-controlled trial of porcine versus synthetic secretin for reducing symptoms of autism. J Am Acad Child Adolesc Psychiatry. 2002 Nov;41(11):1315-21. doi: 10.1097/00004583-200211000-00012. PMID 12410073
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711